CLINICAL TRIAL: NCT03996304
Title: Finnish Health and Early Life Microbiota (HELMi) Longitudinal Birth Cohort
Brief Title: Health and Early Life Microbiota
Acronym: HELMi
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Helsinki (Other)
Collaborators: Business Finland (Other); Valio Ltd (Industry); Finnish Red Cross Blood Service (Other); DuPont Nutrition and Health (Industry); Oriola Corporation (Unknown); Pikkujätti Medical Centre for Children and Youth (Unknown)
Responsible Party: Principal Investigator, Anne Salonen, Principal Investigator, University of Helsinki
Other Study IDs: 263/13/03/03/2015
Record Dates: First submitted 2019-03-26; First posted 2019-06-24 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Child Development; Growth; Allergy; Overweight; Infectious Disease; Noncommunicable Diseases
Keywords: Birth cohort; Intestinal microbiota; Child health
MeSH Terms: conditions — Hypersensitivity; Overweight; Communicable Diseases; Noncommunicable Diseases

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Faecal samples from study infants
  * Faecal samples from parents
  * Buccal swap DNA sample from study infants
  * Breast milk
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this cohort is to identify environmental, lifestyle and genetic factors that modify the human intestinal microbiota development during the first years of life, and to identify early microbiota features that associate to child health and well-being with focus on the development of allergic diseases and overweight.

DETAILED DESCRIPTION:
1055 healthy term infants born in 2016-2018 mainly at the capital region of Finland, and their parents. Fecal samples collected from infants and their parents. Electronic questionnaires on a weekly basis during the first 4 months of life, thereafter less frequently. Focus on diet, well-being and health and social manners. At one-year and at two-years comprehensive questionnaires including development and cognition. Parental stress evaluation included.

ELIGIBILITY:
Inclusion Criteria:

* General population, singleton pregnancy, at least one parent Finnish speaking
* Willingness and ability of parents to consent for 2 year follow-up involving frequent electronic questionnaires and freezing of faecal samples at home
* Infant born on gestational weeks 37-42 without known congenital defects

Exclusion Criteria

* Preterm birth
* Severe birth defect
* Parents fail to activate the online questionnaires

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The cohort consists of 1055 healthy term infants born in 2016-2018 mainly at the capital region of Finland, and their parents.
Sampling Method: Non-Probability Sample
Enrollment: 1055 (Actual)
Dates: Start 2016-02-26 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Longitudinal change of intestinal microbiota in early life | From 3 weeks to 2 years after birth
  Developmental trajectory of the intestinal microbiota, assessed with 16S rRNA gene amplicon and shotgun sequencing of fecal DNA to determine the changes in the intestinal microbiota composition, diversity and functionality from week 3 to weeks 6,9,12 and months 6,9,12,18 and 24 after birth.

SECONDARY OUTCOMES:
Number of children with asthma | At 2 years
  Specialist/Physician-diagnosed asthma.
Number of children with allergic disease | At 2 years
  Specialist/Physician-diagnosed wheeze, eczema/atopic dermatitis, allergic rhinitis, food allergy or atopy.
Number of respiratory tract infection episodes | From birth to 2 years of age
  Number of physician-diagnosed respiratory track infections.
Weight | At 6,12,18 and 24 months after birth
  Weight in kilograms.
Growth | At 6,12,18 and 24 months after birth
  Height in centimeters.
Child development | At 18 and 24 months after birth
  By means of questionnaires and, on a randomly selected group of study subjects, developmental testing to assess cognitive, motor, socio-emotional and verbal development.

CONTACTS AND LOCATIONS:
Overall Officials: Willem M de Vos, Professor, Study Director — University of Helsinki; Anne Salonen, PhD, Principal Investigator — University of Helsinki; Kaija-Leena Kolho, Professor, Principal Investigator — University of Helsinki
Locations (1):
- Human Microbiome Research Program, Faculty of Medicine, University of Helsinki, Helsinki, Finland

REFERENCES:
- [Derived] Korpela K, Kallio S, Salonen A, Hero M, Kukkonen AK, Miettinen PJ, Savilahti E, Kohva E, Kariola L, Suutela M, Tarkkanen A, de Vos WM, Raivio T, Kuitunen M. Gut microbiota develop towards an adult profile in a sex-specific manner during puberty. Sci Rep. 2021 Dec 2;11(1):23297. doi: 10.1038/s41598-021-02375-z. PMID 34857814
- [Derived] Korpela K, Dikareva E, Hanski E, Kolho KL, de Vos WM, Salonen A. Cohort profile: Finnish Health and Early Life Microbiota (HELMi) longitudinal birth cohort. BMJ Open. 2019 Jun 27;9(6):e028500. doi: 10.1136/bmjopen-2018-028500. PMID 31253623